CLINICAL TRIAL: NCT01025440
Title: An Investigation to Test the Efficacy of a Novel CPAP Concept to Reduce the Apnea Hypopnea Index of Patients With Obstructive Sleep Apnea
Brief Title: An Investigation to Test the Efficacy of the High Flow (HF) Continuous Positive Airway Pressure (CPAP) in Patients With Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Collaborators: Helios Klinik Ambrock (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FPHC LP-CPAP09-01
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPAP (Active Comparator): Continuous Positive Airway Pressure (CPAP) is the gold-standard treatment for OSA. CPAP mechanically splints the upper airway open during sleep to prevent collapse and in this way ameliorates OSA.
  Dose: The CPAP pressure will be set to the individual subject's therapeutic pressure -as determined by PSG on Night 2.
  Duration: 1 night - the duration of the subject's sleep period (minimum of 3 hrs of sleep required)
  Interventions: Device: Continuous Positive Airway Pressure
- HFCPAP (Active Comparator): Continuous Positive Airway Pressure (CPAP) is the gold-standard treatment for OSA. CPAP mechanically splints the upper airway open during sleep to prevent collapse and in this way ameliorates OSA.
  Dose: During HF CPAP 35 L/min wil be administered.
  Duration: 1 night - the duration of the subject's sleep period (minimum of 3 hrs of sleep required)
  Interventions: Device: Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — Continuous Positive Airway Pressure (CPAP) Dose: A flow (35 L/min) or pressure (btw 4 and 20 cmH20 -individual to each subject) is set on the device.
  Duration: 1 night - the duration of the subject's sleep period (minimum of 3 hrs of sleep required)
  Duration:
  Other Names: Positive airway pressure

SUMMARY:
Phase One:

High Flow (HF) CPAP (HF-CPAP) Titration:

Participants will attend the sleep lab to undergo a comprehensive split-night respiratory PSG. Each participant will be randomized to one of 20 L/min or 35 L/min of CPAP for the first half of the night and swapped to the alternate flow rate for the second half o the night.

At the completion of night 3 participants will be categorized as responders or non-responders. Only responders will continue to Phase 2 of the investigation.

Phase Two:

HF-CPAP compared with CPAP:

Participants will attend the sleep lab to undergo a comprehensive overnight respiratory PSG. Each participant will be randomized to HF-CPAP at a flow rate of 35 L/min or to conventional CPAP at their therapeutic pressure. They will spend the entire night on this treatment arm. Thew following night participants will undergo the alternative treatment arm for the duration of the night.

DETAILED DESCRIPTION:
Each patient will complete a clinical consultation followed by admission to the HELIOS Klinik Hagen-Ambrock facility to undergo routine assessment, diagnosis and CPAP titration (if necessary) of OSA. This will be performed according to the routine clinical care procedures and protocols of the site. The eligibility of each participant will be established during these routine clinical care nights. After night 2 eligible participants will be offered participation in the investigation.

Phase One:

Night 1 (Routine Clinical Care) Participants will attend the HELIOS Klinik Hagen-Ambrock sleep lab to undergo a comprehensive overnight diagnostic PSG, in order to establish the existence and severity of OSA. If the participant has

1. a positive diagnosis of OSA with an AHI > 15 events/hr and
2. ≥ 90% of all events are Hypopneas they will be eligible to progress to Night 3. Night 2 (Routine Clinical Care) Participants will attend the HELIOS Klinik Hagen-Ambrock sleep lab to undergo a standard CPAP titration, in order to determine their therapeutic CPAP pressure. At this stage, if the participant is eligible, they will be offered participation in the investigation. If potential participants are ineligible or unwilling to participate, they will continue along the routine clinical care path.

Night 3 (Flow Titration) Consented participants will attend the HELIOS Klinik Hagen-Ambrock sleep lab to undergo a comprehensive split-night respiratory PSG.

Each participant will be randomized to one of 20 L/min or 35 L/min of HF-CPAP for the first half of the night. A minimum of three hours on this flow must be recorded on the PSG before participants can be swapped to the alternate flow. Three hours on the alternate flow is also required for this half of the night to be deemed successful.

Responder/Non-responder Determination At the completion of night 3 participants will be categorized as responders or non-responders.

Only responders will continue to Phase 2 of the investigation. A responder is someone who;

1. Achieves a > 50% reduction in AHI and
2. Achieves an RDI < 10 events/hr. Investigation Break Before responders progress to Phase Two participants will be sent home for 1 week. During this time they will be instructed to undertake CPAP treatment. Their CPAP device will be set to their therapeutic pressure which was determined on Night 2.

Phase Two:

Night 4 (HF-CPAP compared with CPAP) Participants will attend the HELIOS Klinik Hagen-Ambrock sleep lab to undergo a comprehensive overnight respiratory PSG.

Each participant will be randomized to OpenCPAP at a flow rate of 35 L/min or to conventional CPAP at their therapeutic pressure. They will spend the entire night on this treatment arm.

Night 5 (HF-CPAP compared with CPAP) Participants will attend the HELIOS Klinik Hagen-Ambrock sleep lab to undergo a comprehensive overnight respiratory PSG.

Participants will be swapped to the alternative treatment arm, either HF-CPAP at a flow rate of 35 L/min or to conventional CPAP at their therapeutic pressure. They will spend the entire night on this treatment. In the morning at completion of the PSG, participants will be asked which treatment Night (4 or 5) they preferred.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years.
* AHI > 15 events per hour and ≥ 90% of events must be Hypopneas.

Exclusion Criteria:

* Any medical condition which contraindicates the use of CPAP or AutoCPAP. See Appendix D for this list.
* Requires supplemental oxygen.
* Unstable cardiovascular disease (untreated or resistant hypertension acceptable).
* Unstable psychiatric disease.
* Other significant sleep disorder.
* Inability to tolerate CPAP due to nasal obstruction or claustrophobia, as determined by the investigation investigator.
* Any known factor or disease that might interfere with treatment compliance, investigation conduct or interpretation of the results such as psychiatric disease, history of non compliance to medical regimens, or unwillingness to comply with investigational requirements.
* Participation in another clinical investigation in the previous month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Efficacy to treat OSA | Nights 3, 4 and 5 (after each PSG)

SECONDARY OUTCOMES:
Sleep Quality | Nights 3, 4 and 5 (after each PSG)
Participant Treatment Preference: HF-CPAP compared with CPAP | Night 5

CONTACTS AND LOCATIONS:
Overall Officials: George Nilius, M.D, Principal Investigator — HELIOS-Klinik Hagen Ambrock
Locations (1):
- HELIOS-Klinik Hagen Ambrock, Ambrocker Weg 60, Hagen, Germany

IPD SHARING:
Plan to Share IPD: Undecided